CLINICAL TRIAL: NCT05231395
Title: Effects of Inspiratory Muscle Training on Oxygen Consumption Muscle Oxygenation and Physical Activity Level in Patients With Post-COVID-19
Brief Title: Effects of Inspiratory Muscle Training in Patients With Post COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gazi University-
Record Dates: First submitted 2022-02-08; First posted 2022-02-09 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: COVID-19; inspiratory muscle training; oxygen consumption; physical activity
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
  Evaluations and interventions will be performed different physiotherapist. In addition, before statistical analysis patients' groups will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training Group (Experimental): Patients in the training group will be performed inspiratory muscle training with the PowerBreathe® (inspiratory muscle training device) device at 50% of the maximal inspiratory pressure.
  Interventions: Other: Inspiratory Muscle Training Group
- Control Group (Sham Comparator): Control group will be given breathing exercises as a home program for 8 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Inspiratory Muscle Training Group — Patients in the training group will receive inspiratory muscle training with the PowerBreathe® (inspiratory muscle training device) at 50% of the maximal inspiratory pressure.
  Patients in the training group inspiratory muscle training will be given 2 sets of 15 minutes a day for a total of 30 minutes/per day or a single session for 30 minutes/week, 7 days/week for a total of 8 weeks.
  Patients in the training group will be given respiratory muscle strength training with a home program 6 days a week under the supervision of a physiotherapist 1 day a week.
  Arms: Inspiratory Muscle Training Group
Other: Control Group — Control group will be given breathing exercises 120 times/day, 7days/week, for 8 weeks as home program.
  Control group will be followed-up by telephone once a week
  Arms: Control Group

SUMMARY:
Coronavirus-2019 (COVID-19) is a new virus that emerged in December 2019 and spread quickly all over the world. Problems such as hypoxia, dyspnea, increased fatigue, decreased exercise capacity and respiratory muscle strength occur in COVID-19 patients.In addition, abnormalities in skeletal muscles due to systemic inflammation, mechanical ventilation, sedation and prolonged bed rest in hospital and intensive care patients cause decreased exercise capacity.

DETAILED DESCRIPTION:
Dyspnea is one of the most common long-term symptoms in COVID-19 patients. It has been determined that dyspnea that persists three and six months after hospital discharge is associated with peak oxygen consumption in hospitalized and discharged COVID-19 patients, while peak oxygen consumption decreases in patients with dyspnea. Inspiratory muscle training may be an effective treatment modality in the treatment of dyspnea in patients with dyspnea after COVID-19. The effects of inspiratory muscle training have been investigated in different lung diseases. In these studies, inspiratory muscle training increased respiratory muscle strength and endurance, exercise capacity, and quality of life, and decreased fatigue and dyspnea.

The aim of this study is to investigate the effects of inspiratory muscle training on oxygen consumption, muscle oxygenation, physical activity level, respiratory muscle strength and endurance, peripheral muscle strength, functional exercise capacity, dyspnea, fatigue and quality of life in patients with COVID-19.

Primary outcome measurement will be oxygen consumption (cardiopulmonary exercise test).

Secondary outcome will be muscle oxygenation (Moxy device), physical activity level (multi sensor activity device), pulmonary function (spirometer), functional exercise capacity (six-minute walk test), respiratory (mouth pressure device) and peripheral muscle (hand-held dynamometer) strength, inspiratory muscle endurance (incremental threshold loading test), functional status (Post-COVID-19 Functional Status Scale), dyspnea (London Chest Daily Living Activity Scale), fatigue (Fatigue Severity Scale) and quality of life (Saint George Respiratory Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75
* Diagnosed with COVID-19
* COVID-19 Polymerase Chain Reaction (PCR) test result negative
* Volunteer to participate in the study

Exclusion Criteria:

* Body mass index >35 kg/m2
* Acute pulmonary exacerbation, acute upper or lower respiratory tract infection
* Aortic stenosis, complex arrhythmia, aortic aneurysm
* Serious neurological, neuromuscular, orthopedic, other systemic diseases or other diseases affecting physical functions
* Cognitive impairment that causes difficulty in understanding and following exercise test instructions
* Participated in a planned exercise program in the last three months
* Bulla formation in the lung
* Uncontrolled hypertension and/or diabetes mellitus, heart failure and cardiovascular disease
* Contraindication for exercise testing and/or exercise training according to the American College of Sports Medicine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Oxygen Consumption | First Day
  Cardiopulmonary Exercises Test

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Second day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria.
Respiratory Muscle Endurance | Second day
  Incremental threshold loading test
Peripheral Muscle Strength | Second day
  Hand held dynamometer
Functional exercise capacity | Second day
  6 minute walking test
Fatigue Severity | First day
  Fatigue Severity Scale (Turkish version) - Fatigue Severity Scale (FSS) is a self-reported questionnaire. FSS evaluates patient's fatigue severity. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Respiratory Associated Quality of Life (respiratory) | First day
  St. George Respiratory Questionnaire (Turkish version) (respiratory) - St. George Respiratory Questionnaire (SGRQ) is a self-reported questionnaire. SGRQ evaluates patients' respiratory disease associated quality of life. This questionnaire includes 2 part (part one is about symptoms (one subsection) and part two is about activity (seven subsection)) and 50 items. Some items scored as Likert scale and others scored as dichotomous (true/false).
Dyspnea | First Time
  London Chest Activity of Daily Living scale (LCADL): LCADL evaluates the limitation to perform activities of daily living by dyspnea and looks at four domains: selfcare, domestic, physical and leisure. It is composed of 15 items, which are scored by the patient as follows: 0 (I do not perform this activity because I never had to do it or it is irrelevant), 1 (I do not feel any breathless when performing this activity), 2 (I feel moderate breathless when performing this activity), 3 (I feel a lot of breathless in doing this activity), 4 (I cannot perform this activity due to breathless and I have no one who can do the activity for me) or 5 (I cannot perform this activity anymore and I need someone to do it for me or help me because of breathless).
Muscle oxygenation | First and second day
  Moxy® monitor
Physical Activity Level | Second Day
  Multi sensor activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, Pt. MSc., Principal Investigator — Gazi University; Ece BAYTOK, Pt. MSc., Principal Investigator — Gazi University; Nilgün YILMAZ DEMİRCİ, Assoc.Prof, Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debeaumont D, Boujibar F, Ferrand-Devouge E, Artaud-Macari E, Tamion F, Gravier FE, Smondack P, Cuvelier A, Muir JF, Alexandre K, Bonnevie T. Cardiopulmonary Exercise Testing to Assess Persistent Symptoms at 6 Months in People With COVID-19 Who Survived Hospitalization: A Pilot Study. Phys Ther. 2021 Jun 1;101(6):pzab099. doi: 10.1093/ptj/pzab099. PMID 33735374
- [Background] Abodonya AM, Abdelbasset WK, Awad EA, Elalfy IE, Salem HA, Elsayed SH. Inspiratory muscle training for recovered COVID-19 patients after weaning from mechanical ventilation: A pilot control clinical study. Medicine (Baltimore). 2021 Apr 2;100(13):e25339. doi: 10.1097/MD.0000000000025339. PMID 33787632
- [Background] Anastasio F, Barbuto S, Scarnecchia E, Cosma P, Fugagnoli A, Rossi G, Parravicini M, Parravicini P. Medium-term impact of COVID-19 on pulmonary function, functional capacity and quality of life. Eur Respir J. 2021 Sep 16;58(3):2004015. doi: 10.1183/13993003.04015-2020. Print 2021 Sep. PMID 33574080
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129